CLINICAL TRIAL: NCT06112808
Title: A Double-Blind, Randomized Clinical Study of the Pharmacokinetics and Safety of BCD-263 and Opdivo® as Monotherapy in Subjects With Advanced Melanoma of the Skin
Brief Title: A Clinical Study of the Pharmacokinetics and Safety of BCD-263 and Opdivo® as Monotherapy in Subjects With Advanced Melanoma of the Skin
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCD-263-1
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Advanced Melanoma
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BCD-263 (Experimental)
  Interventions: Drug: BCD-263
- Opdivo (Active Comparator)
  Interventions: Drug: Opdivo

INTERVENTIONS:
Drug: BCD-263 — BCD-263 at a dose 480 mg administered intravenously every 4 weeks up to 6 cycles
  Other Names: Nivolumab
  Arms: BCD-263
Drug: Opdivo — Opdivo at a dose 480 mg administered intravenously every 4 weeks up to 6 cycles
  Other Names: Nivolumab
  Arms: Opdivo

SUMMARY:
The aim of the study BCD-263-1 is to prove the comparability of the pharmacokinetics and similarity of the safety, immunogenicity and pharmacodynamic profiles of BCD-263 and Opdivo following intravenous administration to subjects with advanced unresectable or metastatic melanoma of the skin. The study will have randomized, double-blind design with parallel assignment.

DETAILED DESCRIPTION:
Following screening, subjects will be randomized to receive either BCD-263 or Opdivo in a 1:1 ratio and enter the main study period.

During the main study period, subjects will receive therapy with BCD-263 or Opdivo, which will be administered intravenously until disease progression or signs of unacceptable toxicity develop (whichever occurs earlier).

At Week 25, after completion of all scheduled procedures subjects in both groups will continue to receive open-label BCD-263 for up to a total of 2 years of therapy, or disease progression, or signs of unacceptable toxicity (whichever occurs first).

Following discontinuation of the study therapy, the subjects will enter a follow-up period, during which data on overall survival will be collected through telephone contacts.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of signing the informed consent form;
2. Body weight 60 to 90 kg.
3. Histologically confirmed melanoma with the following prognostic characteristics:

   * LDH <ULN of local laboratory (enrollment of subjects with LDH <2x ULN of local laboratory is allowed until the number of subjects with LDH >ULN is 30% of the total population of randomized subjects. The Sponsor will inform when enrollment of subjects is limited by LDH level <ULN of the local laboratory).
   * Absence, according to the Investigator, of clinically significant symptoms associated with the tumor.
   * Absence, according to the Investigator, of rapidly progressing metastatic melanoma.
4. Newly diagnosed advanced unresectable (stage III) or metastatic disease (stage IV), or progressive disease during / relapsing after radical treatment.

Exclusion Criteria:

1. Indications for radical treatment (surgery, radiation therapy).
2. Uveal or mucosal melanoma.
3. Previous systemic anticancer therapy for advanced unresectable or metastatic skin melanoma (a history of neoadjuvant or adjuvant therapy is allowed, provided that the therapy was completed at least 12 weeks before randomization).
4. Active CNS metastases and/or carcinomatous meningitis.
5. Previous invasive cancer, excluding diseases treated with potentially curative therapy with no evidence of recurrence for 2 years from the start of this therapy (subjects with radically resected basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, cervical carcinoma in situ of the uterus and other carcinomas in situ may be included).
6. Subjects with severe concomitant disorders, life-threatening acute complications of the primary disease (including massive pleural, pericardial, or peritoneal effusions requiring intervention, pulmonary lymphangitis, bleeding or organ perforation) at the time of signing the informed consent and during the screening period.
7. Concomitant diseases and/or conditions that significantly increase the risk of adverse events (AEs) during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
AUC(0-672) of nivolumab | pre-dose to week 25
  To compare area under the drug concentration-time curve in the time interval from 0 to 672 hours after intravenous administration of BCD-263 and Opdivo

SECONDARY OUTCOMES:
Cmax | week 25
  To compare the maximum concentration of nivolumab after intravenous administration of BCD-263 and Opdivo
AUC(0-∞) | week 25
  To compare area under the drug concentration-time curve in the time interval from 0 to ∞ after intravenous administration of BCD-263 and Opdivo
Tmax | week 25
  To compare time to the maximum concentration of nivolumab after intravenous administration of BCD-263 and Opdivo
T½ | week 25
  To compare half-life period of nivolumab after intravenous administration of BCD-263 and Opdivo
Kel | week 25
  To compare elimination rate constant of nivolumab after intravenous administration of BCD-263 and Opdivo
Vd | week 25
  To compare steady-state volume of distribution of nivolumab after intravenous administration of BCD-263 and Opdivo
Cl | week 25
  To compare total clearance of nivolumab after intravenous administration of BCD-263 and Opdivo
Ceoi | week 25
  To compare plasma concentration at the and of infusion of nivolumab after intravenous administration of BCD-263 and Opdivo
Ctrough | week 25
  To compare trough concentration at the and of infusion of nivolumab after intravenous administration of BCD-263 and Opdivo
Safety assessment | week 25
  The subjects will undergo the vital sign assessment, physical and instrumental examination, sampling for complete blood count, blood chemistry, thyroid hormone tests, and urinalysis, as well as assessment of the presence and characteristics of adverse events to assess the safety of the investigational product
Immunogenicity assessment | week 25
  Proportion of subjects with binding and/or neutralizing antibodies to nivolumab
Pharmacodynamics assessment | week 25
  Occupancy of PD-1 receptors on CD4+ and CD8+ peripheral blood lymphocytes
Efficacy assessment: ORR | week 25
  To compare overall response rate according to RECIST 1.1 and iRECIST criteria after administration of BCD-263 or Opdivo
Efficacy assessment: PFS | week 25
  To compare progression-free survival according to RECIST 1.1 and iRECIST criteria after administration of BCD-263 or Opdivo
Efficacy assessment: overall survival | week 25
  To compare overall survival according to RECIST 1.1 and iRECIST criteria after administration of BCD-263 or Opdivo
Efficacy assessment: DCR | week 25
  To compare disease control rate according to RECIST 1.1 and iRECIST criteria after administration of BCD-263 or Opdivo
Efficacy assessment: time to response | week 25
  To compare time to response according to RECIST 1.1 and iRECIST criteria after administration of BCD-263 or Opdivo
Efficacy assessment: duration of response | week 25
  To compare duration of response according to RECIST 1.1 and iRECIST criteria after administration of BCD-263 or Opdivo

CONTACTS AND LOCATIONS:
Overall Officials: Arina V Zinkina-Orikhan, Study Director — Director of Clinical Development Department, BIOCAD
Locations (30):
- Belarus (2):
  - Healthcare Institution "Minsk City Clinical Cancer Center", Minsk
  - State Institution "Republic Scientific and Practical Centre for Oncology and Medical Radiology Named after N.N.Aleksandrov", Minsk
- Russia (28):
  - Chelyabinsk Regional Clinical Center for Oncology and Nuclear Medicine, Chelyabinsk, Chelyabinsk Oblast
  - JSC "Modern Medical Technologies", Saint Petersburg, Sankt-Peterburg
  - LLC "New Clinic", Pyatigorsk, Stavropol Kray
  - State Budgetary Institution of Healthcare of the Arkhangelsk Region "Severodvinsk City Hospital №2 of Emergency", Arkhangelsk
  - Regional State Budgetary Healthcare Institution "Altai Regional Oncological Dispensary", Barnaul
  - Federal State Educational Institution of Higher Education "Baltic Federal University Named after Immanuel Kant", Kaliningrad
  - Limited Liability Company "Ars Medica Centre", Kaliningrad
  - State Budgetary Healthcare Institution of Kaluga Region "Kaluga Region Clinical Oncological Dispensary", Kaluga
  - State Autonomous Health Institution "Republican Clinical Oncology Dispensary of the Ministry of Health of the Republic of Tatarstan named after Professor M.Z. Sigal", Kazan'
  - Regional State Budgetary of Healthcare Insti-tution "Kostroma Clinical Oncology Dispensary", Kostroma
  - "Russian Cancer Research Center named after N.N. Blokhin "of the Ministry of Health of the Russian Federation, Moscow
  - JSC "Medsi Group", Moscow
  - Moscow City Oncology Hospital No. 62, Moscow
  - State budgetary health care institution of the city of Moscow "City Clinical Oncology Hospital No. 1 of the Department of Health of the City of Moscow", Moscow
  - State Budgetary Healthcare Institution "Moscow Clinical Scientific Center funded by Moscow Health Department" (SBHI MCSC MHD), Moscow
  - Nizhny Novgorod Region State Budgetary Healthcare Institution "Nizhny Novgorod Regional Clinical Oncological Dispensary", Nizhny Novgorod
  - State Budgetary Healthcare Institution of Novosibirsk Region "Novosibirsk Region Clinical Oncological Dispensary", Novosibirsk
  - State budget healthcare institution Omsk region "Clinical Oncology Dispensary", Omsk
  - Private healthcare institution "Clinical hospital "RZD-Medicine" of the city of Saint Petersburg", Saint Petersburg
  - "Saint Petersburg Clinical Research and Practice Center for Specialized Medical Care (Oncology)", Saint Petersburg
  - Federal State Budgetary Institution "N.N. Petrov Research Institute of Oncology" of the Ministry of Healthcare of the Russian Federation, Saint Petersburg
  - Limited Liability Company "Oncological Research Center", Saint Petersburg
  - Private Medical Institution Evromedservis, Saint Petersburg
  - State-financed Health Institution "Samara Region Clinical Oncology Dispensary", Samara
  - Federal State Educational Institution of Higher Professional Education "Mordovia State University N.P. Ogareva ", Saransk
  - Limited Liability Company "Nebbiolo", Tomsk
  - Republican Clinical Oncology Dispensary of Ministry of Health republic Bashkortostan, Ufa
  - State Health Care Institution "Volgograd Regional Clinical Oncology Dispensary № 1", Volgograd

IPD SHARING:
Plan to Share IPD: No